CLINICAL TRIAL: NCT02913521
Title: A Double-Blind, Randomized, Placebo-Controlled, Parallel Group, Three-Arm, Multi-Site Study to Evaluate the Clinical Equivalence of Diclofenac Sodium Topical Gel 1% (Hi-Tech Pharmacal Co., Inc.) With Voltaren® Gel (Diclofenac Sodium Topical Gel) 1% (Novartis) in Patients With Osteoarthritis of the Knee
Brief Title: Bioequivalence Study With Clinical Endpoint for Diclofenac Sodium Topical Gel 1%
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Akorn, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P130021
Record Dates: First submitted 2016-09-22; First posted 2016-09-23 (Estimated); Results first posted 2021-02-26 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-01

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Diclofenac Sodium Gel 1% (Experimental): Apply 4 g of gel to the knee four times a day
  Interventions: Drug: Diclofenac Sodium Gel 1%
- Voltaren Gel (Active Comparator): Apply 4 g of gel to the knee four times a day
  Interventions: Drug: Voltaren Gel
- Placebo (Placebo Comparator): Apply 4 g of gel to the knee four times a day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Diclofenac Sodium Gel 1%
  Arms: Diclofenac Sodium Gel 1%
Drug: Voltaren Gel
  Arms: Voltaren Gel
Drug: Placebo
  Arms: Placebo

SUMMARY:
A Double-Blind, Randomized, Placebo-Controlled, Parallel Group, Three-Arm, Multi-Site Study to Evaluate the Therapeutic Equivalence of Diclofenac Sodium Topical Gel 1% (Hi-Tech Pharmacal Co., Inc.) With Voltaren® Gel (Diclofenac Sodium Topical Gel) 1% (Novartis) in Patients With Osteoarthritis of the Knee

ELIGIBILITY:
Inclusion Criteria:

1. Ambulatory male and non-pregnant females 35 years and older diagnosed with osteoarthritis according to the American College of Rheumatology Criteria (ACR) in one knee. Target knee is the one with higher level of pain.

   ACR Criteria includes: Knee Pain and at least 3 of the following: age ≥ 50, stiffness lasting < 30 mins, bony tenderness, crepitus, bony enlargement, and no palpable warmth.
2. Symptom onset of > 6 Months prior to Screening for the target knee.
3. If female and of child-bearing potential, prepare to abstain from sexual intercourse or use a reliable method of contraception during the study (e.g., IUD, oral, transdermal, injected, implanted hormonal contraceptives or condom + spermicide).
4. Periarticular knee pain due to osteoarthritis (not bursitis, tendonitis etc.) that required the use of oral or topical treatments (e.g., NSAIDs or acetaminophen).
5. Radiograph of the target knee within the previous year with a Grade 1, 2 or 3 disease based upon the Kellgren-Lawrence disease severity scale.
6. After a minimum of 7-day wash out of all pain medication has Baseline pain on movement score of ≥ 50mm on a 0-100-mm Visual Analogue Scale for the target knee.
7. After a minimum of 7-day wash out of all pain medication has Baseline WOMAC Pain sub scale of ≥ 9 on a 5 question, 5 point (0 to 4) Likert scale for the target knee.
8. Willing and able to use only acetaminophen as rescue medication.
9. Willing and able to comply with the study requirements.

Exclusion Criteria:

1. Females who are pregnant, breast feeding, or planning a pregnancy.
2. Radiograph of the target knee within the previous year with a Grade 4 score on the Kellgren-Lawrence disease severity scale.
3. History of osteoarthritis in the contralateral knee requiring medication (OTC or prescription) within 12 months of screening.
4. After a minimum of 7-day wash out of all pain medication has Baseline pain on movement score of ≥ 20mm on a 0-100-mm Visual Analogue Scale for the contralateral knee immediately prior to randomization.
5. Known history of secondary osteoarthritis (e.g. congenital, traumatic, gouty arthritis) of the knee or rheumatoid arthritis.
6. Known history of other chronic inflammatory diseases, (e.g., colitis) or fibromyalgia during last 5 years. Patients whose disease was diagnosed at least 5 (five) years prior to screening visit and have had no known disease activity (i.e., no disease related complaints nor disease treatment prescribed) since then may enter into the study.
7. History of asthma, hypertension, myocardial infarction, thrombotic events, stroke, congestive heart failure, impaired renal function or liver disease. Patients who have had high blood pressure measured at least 2 (two) years prior to screening visit and have had no disease activity (i.e., no record of hypertension or anti-hypertensive treatment prescribed) for at least 2 (two) years prior to screening visit may enter into the study.
8. History of coronary artery bypass graft within 6 months of screening.
9. Concomitant acetylsalicylic acid therapy other than a stable low dose used for cardiac prophylaxis (max. 162 mg daily) taken for at least 3 months prior to enrollment and maintained throughout the duration of the study.
10. Use of warfarin or other anticoagulant therapy within 30 days of screening.
11. Use of ACE inhibitors, cyclosporine, diuretics, lithium or methotrexate, within 30 days of screening or during the study.
12. Known history of gastrointestinal bleeding or peptic ulcer disease.
13. Abnormal screening clinical laboratory evaluations which the Investigator deems clinically significant.
14. Known allergy to aspirin or NSAIDs.
15. Skin lesions or wounds in the affected area.
16. Significant (requiring surgery) injury or major knee surgery to either knee within six months prior to screening.
17. Transaminase levels that are more than two times the upper limit of the normal range at screening.
18. Any other acute or chronic illness that in the opinion of the investigator could compromise the integrity of study data or place the Patient at risk by participating in the study.
19. Concomitant use of corticosteroids (any formulation) or use within 30 days of study randomization.
20. Receipt of any drug as part of a research study within 30 days prior to screening.
21. Previous randomization into this study.
22. Known allergy (hypersensitivity) to acetaminophen.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 934 (Actual)
Dates: Start 2015-06; Primary Completion 2016-04 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kalev Kask, Ph.D., Study Director — EGeen International Inc.
Locations (50):
- Estonia (12):
  - Vee Family Doctor's Center OY, Paide
  - OU Mai Perearstid, Pärnu
  - East Tallinn Central Hospital, Tallinn
  - West Tallinn Central Hospital, Tallinn
  - Medicum Ltd., Tallinn
  - Linna Health Cerntre, Tallinn
  - Linnamoisa Perearstikeskus, Tallinn
  - OU Perearstikeskus Remedium, Tallinn
  - Pirita Family Doctors Centre, Tallinn
  - Orthopaedic and Clinical Research Center, Tartu
  - Dr.Monika Vask Ltd., Tartu
  - Ltd. Elli Kahar, Tartu
- Latvia (4):
  - Association of Health Centres, Medical Centre "OLVI", Daugavpils
  - D.Saulites-Kandevicas private practice, Liepāja
  - SIS Klinika ALma, Riga
  - Health Center 4, Riga
- Lithuania (5):
  - InMedica, Kaunas
  - JSC Vita Longa, Kaunas
  - JSC Saules seimos medicinos centras, Kaunas
  - JSC Mano Seimos Gydytojas, Klaipėda
  - Private Doctor Family Clinic JSc Ausveja, Vilnius
- Poland (11):
  - Medical Chamber in Warsaw Nr 5718455, Warsaw, Masovian Voivodeship
  - CERMED, Bialystok
  - ClinicMed Badurski i Wspolnicy Spolka Jawna, Bialystok
  - St. Luke's hospital in Bielsko-Biala, Bielsko-Biala
  - Private medical practice Jacek Niski, Częstochowa
  - Niepubliczny Zaklad Opieki Zdrowotnej ORTMED sp. z o.o., Lodz
  - Clinical Best Solutions, Lublin
  - MEDICOME Sp. z o.o., Oświęcim
  - ZOZ w Olawie, Oława
  - Centrum Medyczne Luxmed, Przezmierowo, Poznan
  - "REUMA TIKA- Centrnrn Reurnatologii" NZOZ, Warsaw
- Romania (9):
  - Spiratul Judetean de Urgenta Bacau, Bacau
  - Spital Judetean De Urgenta Bacau, Bacau
  - Duo Medical, Bucharest
  - S.C. lanuli Med Consult Str Intr Lt. Dumitru Lemnea, Bucharest
  - Dr Ion Stoia Rheumatology Center, Bucharest
  - Emergency County Hospital SF Gheorghe, Bucharest
  - RK Medcenter SRL, Iași
  - S.C. Clinica Somesan, Mărăști
  - Ploiești Municipal Hospital, Ploieşti
- Ukraine (9):
  - Communal Institution "Cherkasy Regional Hospital of Cherkasy Regional Council", Cherkasy
  - State Institution "Ukrainian State Scientific and Research Institute of Medical and Social Problems of Disability of the Ministry of Health of Ukraine, Dnipropetrovsk
  - State Institution "Professor M.I. Sytenko Institute of Spine and Joint Patholo of the National Academ of Medical Sciences of Ukraine, Kharkiv
  - Communal Institution of Kyiv Regional Council "Kyiv Regional Clinical Hospital", Kyiv
  - State Institution D.F.Chebotariov Institute of Gerontology of NAMS of Ukraine, Kyiv
  - State Institution D.F.Chebotariov Institute ofGerontolo!.!v ofNAMS of Ukraine - Dept of Age related changes to Muscoskeletal system, Kyiv
  - Communal Institution of.Lviv Regional Council "Yu. Lypa Lviv Regional Hospital of Disabled War Veterans and Former Political Prisoners", Lviv
  - Odesa Regional Clinical Hospital, Odesa
  - MI Pyogrov Vinnystya Regional Clinical Hospital, Vinnytsia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Diclofenac Sodium Gel 1%: Apply 4 g of gel to the knee four times a day
  Diclofenac Sodium Gel 1%
- Voltaren Gel: Apply 4 g of gel to the knee four times a day
  Voltaren Gel
- Placebo: Apply 4 g of gel to the knee four times a day
  Placebo
Period: Overall Study
Arm/Group | Diclofenac Sodium Gel 1% | Voltaren Gel | Placebo
Started | 316 | 312 | 306
Completed | 263 | 262 | 261
Not Completed | 53 | 50 | 45

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Diclofenac Sodium Gel 1% | Voltaren Gel | Placebo | Total
Number analyzed (Participants) | 263 | 262 | 261 | 786
Age, Continuous [Mean (Standard Deviation); unit: year] — Population: ITT population described below
  year | 58 (10.3) | 58 (11.1) | 57 (10.8) | 57.3 (11)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: ITT population
  Participants
    Female | 200 | 193 | 190 | 583
    Male | 63 | 69 | 71 | 203

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline to Week 8 in WOMAC Pain Scale, Bioequivalence of Test to Reference.
Description: WOMAC = Western Ontario and McMaster Universities Arthritis Index. The higher number is more pain. Change from baseline to Week 8 as indicated in the title. Scale is 5 questions with a scale of 0-4, higher number is more pain. Therefore, if you have 5 questions and the max score for each is 4, the maximum number on the scale is 20 (5 questions x 4 units on the scale = 20).
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Diclofenac Sodium Gel 1% | Voltaren Gel | Placebo
Number analyzed (Participants) | 258 | 255 | 257
units on a scale | 6.8 (2.1) | 6.7 (2.3) | 5.9 (2.4)

2. Secondary Outcome: An Evaluation to Determine Superiority of Test and Reference Against Placebo in the Mean Change From Baseline to Week 8 in the Total WOMAC Pain Score.
Description: as for outcome 1
Time Frame: 8 weeks
Population: mITT
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Diclofenac Sodium Gel 1% | Voltaren Gel | Placebo
Number analyzed (Participants) | 263 | 262 | 261
units on a scale | 6.8 (1.9) | 6.6 (2.0) | 5.9 (2.1)

3. Secondary Outcome: Incidences of Treatment Emergent Adverse Events
Time Frame: 8 weeks
Reporting Status: Not Posted

4. Secondary Outcome: Incidences of Abnormal Vital Signs
Time Frame: 8 weeks
Reporting Status: Not Posted

5. Secondary Outcome: Clinically Significant Changes From Baseline in Physical Examination Results
Time Frame: 8 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Diclofenac Sodium Gel 1% | Voltaren Gel | Placebo
All-Cause Mortality (participants affected / at risk) | 0/316 | 0/312 | 0/306
Serious Adverse Events (participants affected / at risk) | 0/316 | 0/312 | 0/306
Other Adverse Events (participants affected / at risk) | 30/316 | 24/312 | 20/306
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Diclofenac Sodium Gel 1% (N=316) | Voltaren Gel (N=312) | Placebo (N=306)
application site reaction (Skin and subcutaneous tissue disorders) | 6 (316) | 4 (312) | 3 (306)
General disorders, muscle/skeletal, and nervous system (Investigations) | 24 (316) | 20 (312) | 17 (306)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-21): https://cdn.clinicaltrials.gov/large-docs/21/NCT02913521/Prot_SAP_000.pdf